CLINICAL TRIAL: NCT06139731
Title: Changes in Function of the Upper Limb With Physiotherapy for Acute Burns: a Pilot Study
Brief Title: Changes in Function of the Upper Limb With Physiotherapy
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Brigita Siparyte-Sinkeviciene, Brigita Siparyte-Sinkeviciene, Lithuanian University of Health Sciences
Other Study IDs: Brigita Siparyte-Sinkeviciene
Record Dates: First submitted 2023-10-03; First posted 2023-11-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Burn of Upper Limb, Except Wrist and Hand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This paper describes a pilot clinical study designed to compare changes in ROM, muscle strength and functional recovery of the upper limb during the inpatient treatment period of burn injury.

DETAILED DESCRIPTION:
Patients with burns can face challenges throughout their recovery, including contractures and a reduced range of motion (ROM) in the upper limb (UL), upper and lower limb impairment. Restoring range of motion, muscle strength, and mobility is essential to reduce scarring formation and contractures. The study included 17 patients with unilateral or bilateral superficial, deep partial and full thickness burns to the upper limbs, with or without burns to the upper body, covering 10% or more of the total body surface area

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-69 years
* had burns on the upper limb(s) with or without burns on the upper body
* burns involving ≥ 10% total body surface area (TBSA) with the presence of deep partial thickness or full thickness burns
* who agreed to take part in the study

Exclusion Criteria:

* inability to perform or understand tests
* other injuries (fractures, brain injury)
* central and peripheral nervous system disorders
* amputation
* with burns on the head, hands, feet, and genital area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were invited to participate in the study when they came to the Department of Plastic and Reconstructive Surgery, the Kaunas Clinics, Lithuanian University of Health Sciences, for treatment of burns to the upper limb(s) or upper body. Data for this analysis were collected in 2020-2022.
Sampling Method: Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Upper limb range of motion | Day 0, 7,14,21, 28, 35, more 35 days
  A range of motion assessment evaluates the mobility of the injured joint and assesses the limitations of the range of motion.
Upper limb muscle strength | Day 0,14,35, more than 35 days
  Assessing muscle strength helps determine how much muscle strength will be lost as a patient heals from a burn injury.
Pain intensity | Day 0, 7,14,21, 28, 35, more than 35 days
  The pain rate scale assesses the intensity of pain. A higher score indicates a higher level of pain.
Activities of daily living | Day 0,14,35, more than 35 days
  Assessment of daily activity assesses the limitations of your daily activities. Higher scores associated with greater independence in daily activities.
Functional recovery of the upper limbs | Day 0,14,35, more than 35 days
  Assesses impairment and activity limitation, as well as a restriction of leisure and work activities due to upper limb dysfunction. A higher score indicates a higher degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Rytis Rimdeika, Prof, Principal Investigator — Lithuania LUHS hospital Kaunas Clinics, Department of Plastic and Reconstructive Surgery
Locations (1):
- Brigita Siparytė-Sinkevičienė, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided